CLINICAL TRIAL: NCT05490433
Title: A Prospective Multicenter Randomized Clinical Trial: Robot-assisted vs. Open Nipple-sparing Mastectomy With Immediate Breast Reconstruction (ROM) Trial
Brief Title: Robot-assisted vs. Open Nipple-sparing Mastectomy With Immediate Breast Reconstruction
Acronym: ROM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2022-0600
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Classified as TNM Stage 0-IIIa
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: RNSM and CNSM procedures are systematic at 1:1 ratio after obtaining consent forms for research participation and checking criteria for exclusion from selection It is randomly assigned from the award. The patient is subjected to a single blind examination so that the surgical method is unknown before surgery.
  Reconstruction methods after resection are discussed with breast and/or plastic surgeons
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robot assisted nipple sparing mastectomy(RNSM) (Experimental): Robotic nipple sparing mastectomy, robotic mastectomy, hybrid robotic nipple sparing mastectomy, robotic nipple mammary complex and skin sparing mastectomy, robot nipple sparing mastectomy
  Interventions: Procedure: Robot-assisted Nipple-Sparing Mastectomy (RNSM)
- Conventional nipple sparing mastectomy(CNSM) (Active Comparator): Total mastectomy, mastectomy, nipple sparing mastectomy, skin sparing mastectomy, nipple sparing breast resection, open nipple sparing mastectomy, general nipple sparing Mammastectomy, an open-window nipple sparing mastectomy
  Interventions: Procedure: Conventional nipple sparing mastectomy(CNSM)

INTERVENTIONS:
Procedure: Robot-assisted Nipple-Sparing Mastectomy (RNSM) — Patients undergoing robot-assisted nipple-sparing mastectomy (RNSM) with immediate breast reconstruction (IBR) will be enrolled in this group. RNSM will be performed using robotic surgical platforms, including the da Vinci S, Si, X, Xi, and SP systems. The procedure will be conducted through an axillary or lateral chest wall incision.
  During surgery, posterior areolar tissue sampling for frozen section biopsy will be recommended. If suspicious lesions are detected at the superficial or posterior margins, frozen section biopsy of those lesions will also be performed. When tumor involvement of the nipple-areola complex (NAC), superficial margin, or posterior margin is confirmed by frozen section biopsy, additional resection including the skin and NAC, or postoperative radiotherapy, will be considered.
  Arms: robot assisted nipple sparing mastectomy(RNSM)
Procedure: Conventional nipple sparing mastectomy(CNSM) — Patients who undergo conventional nipple-sparing mastectomy (CNSM) with immediate breast reconstruction (IBR) will be enrolled in this group. CNSM is performed without the use of robotic or endoscopic surgical systems, and all types of skin incisions are permitted.
  During surgery, posterior areolar tissue sampling for frozen section biopsy is recommended. If suspicious lesions suggesting tumor involvement are identified at the superficial or posterior margins, frozen section biopsy should also be performed. When frozen section biopsy confirms tumor involvement of the nipple-areola complex (NAC), superficial margin, or posterior margin, additional excision including the skin and NAC, or postoperative radiotherapy, will be considered.
  Arms: Conventional nipple sparing mastectomy(CNSM)

SUMMARY:
Research Purpose The present study is designed to generate the strongest evidence available on the role of robotic surgical systems in breast cancer surgery and to elucidate the clinical value of immediate breast reconstruction (IBR) conducted in conjunction with robot-assisted nipple-sparing mastectomy (RNSM).

Study Design Overview This study is a prospective, multicenter, randomized clinical trial (ROM Trial) designed to compare the oncologic outcomes of robot-assisted nipple-sparing mastectomy (RNSM) with conventional nipple-sparing mastectomy (CNSM), which includes both traditional and open-chest approaches. Previous retrospective studies of robot-assisted endoscopic surgery have suggested a short learning curve, demonstrating technical feasibility and reproducibility even for less experienced surgeons. However, the absence of rigorously designed randomized clinical trials remains a major global barrier to the broader adoption of robotic breast surgery.

In the ROM Trial, eligible patients who provide written informed consent will be randomly assigned in a 1:1 ratio to undergo either RNSM or CNSM. Participants will be blinded to group allocation until the day of surgery (single-blind design). Immediate breast reconstruction (IBR) will be performed in all patients, with the reconstruction method determined in consultation with the breast and/or plastic surgeon following mastectomy.

DETAILED DESCRIPTION:
Background Robot-assisted nipple-sparing mastectomy (RNSM) has emerged as an approach for both breast cancer treatment and risk-reducing mastectomy in women carrying high-risk pathogenic variants. Although several studies have reported that RNSM is a feasible procedure, concerns remain that it is performed only by a small number of specialized surgeons, and data on oncologic outcomes and patient-reported outcomes (PROs) remain limited. Recently, the United States Food and Drug Administration and several expert surgeons have cautioned that robotic breast surgery should be performed only by highly trained specialists, and that the benefits, risks, and alternative treatment options must be thoroughly discussed with patients to ensure fully informed decision-making.

To promote the safe and standardized application of RNSM, the Korea Robot-Endoscopy Minimal Access Breast Surgery Study Group (KoREa-BSG) was established with the mission to evaluate, standardize, and disseminate this advanced surgical technique.

Study Design We designed a prospective, multicenter, randomized clinical trial (Robot vs. Open Nipple-sparing Mastectomy Trial; ROM Trial) to evaluate the oncologic outcomes of RNSM with immediate breast reconstruction (IBR), compared with conventional open nipple-sparing mastectomy (CNSM) with IBR.

Previous retrospective studies on robot-assisted endoscopic breast surgery have demonstrated a short learning curve, suggesting that the technique is feasible and reproducible even for less experienced surgeons. However, the absence of rigorously designed randomized controlled trials has been a major limitation in expanding the global adoption of robotic breast surgery. The ROM Trial was therefore established to address this unmet need.

Data Collection Clinical and pathological data to be collected include: height, weight, breast volume/weight, age, germline likely pathogenic/pathogenic mutation status, affected breast, bilaterality, breast ptosis, tumor size, TNM stage, histologic grade, histologic type, estrogen receptor (ER), progesterone receptor (PR), human epidermal growth factor receptor 2 (HER2), Ki-67 index, nipple involvement, neoadjuvant/adjuvant treatment status, postoperative complications (Clavien-Dindo classification), operative time, margin involvement, postoperative drainage amount/duration, risk-reducing mastectomy (RRM) status, reconstruction type, recurrence status, healthcare cost data, and follow-up information.

Patient Satisfaction Assessment Between 3 and 12 months (±30 days) after the final surgery, patients will be surveyed using the validated Korean version of the BREAST-Q questionnaire to evaluate satisfaction with surgery.

Cost-Effectiveness Assessment (Optional) Cost-effectiveness according to surgical method will be evaluated between 3 and 12 months (±30 days) after the final surgery, using the Korean version of the EuroQol 5-Dimension (EQ-5D) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (≥19 years) scheduled to undergo therapeutic mastectomy for breast cancer who desire immediate breast reconstruction (IBR).
* Breast cancer classified as clinical TNM stage 0 to IIIA, based on preoperative evaluation according to the 8th edition of the AJCC anatomic staging system.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* Patients scheduled for breast-conserving surgery or deemed ineligible for immediate breast reconstruction (IBR).
* Clinical evidence of nipple or skin involvement on preoperative evaluation.

  * Pregnant or breastfeeding women.
  * Tumors consisting exclusively of lobular carcinoma in situ (LCIS).
  * Paget's disease of the breast.
  * Inflammatory breast cancer.
  * Male breast cancer.
  * Clinical stage IIIB-IV disease on preoperative evaluation.
  * breast size equal to or larger than cup E
  * History of breast cancer or bilateral breast cancer (including metachronous or synchronous disease).
  * History of non-breast malignancy, with the exception of non-melanoma skin cancer or papillary/follicular thyroid carcinoma.
  * Special histologic subtypes of breast tumors (e.g., phyllodes tumor, sarcoma, lymphoma).
  * Age >70 years.
  * American Society of Anesthesiologists (ASA) physical status classification grade ≥4.
  * Inability to provide informed consent.
  * History of prior chest radiotherapy.
  * Patients who have not undergone preoperative testing for hepatitis B virus (HBV), hepatitis C virus (HCV), and human immunodeficiency virus (HIV), which is required for liability insurance coverage.

Ages: 19 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 790 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2032-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
5-year disease-free survival rate(DFS) | The DFS period is calculated from the date of surgery to the time of the first event, or censored at the date of last follow-up if no event is reported.
  From the date of surgery to the first qualifying event, or censored at the date of last follow-up if no event occurs
  * Events: local/regional/distant recurrence, contralateral breast cancer, or all-cause mortality.
  * Local recurrence: recurrence in the ipsilateral breast or chest muscles, ipsilateral chest wall, or nipple-areola complex (NAC).
  * Regional recurrence: recurrence in the ipsilateral axillary lymph nodes, ipsilateral infra/supraclavicular lymph nodes, or ipsilateral internal mammary lymph nodes.
  * intraepithelial carcinoma is included as an event for local recurrence and contralateral breast cancer.
  * patients without an event are censored at the last known disease assessment.
  Statistical analysis (non-inferiority)
  * DFS will be analyzed using a Cox proportional hazards model stratified by institution and clinical stage.
  * The hazard ratio (HR) for RNSM vs CNSM and its 95% confidence interval (CI) will be estimated.

SECONDARY OUTCOMES:
5-Year Overall Survival (OS) | secondary outcome is calculated from the date of surgery to the time the first event occurs, or if the event is not reported on the last follow-up date.(After 5 years of follow-up observation of subject registration)
  Events for OS are defined as death from any cause. OS time will be calculated in months from the date of surgery to the date of the event.
5-Year Breast Cancer-Specific Survival (BCSS) | secondary outcome is calculated from the date of surgery to the time the first event occurs, or if the event is not reported on the last follow-up date.(After 5 years of follow-up observation of subject registration)
  Events for BCSS include death attributable to breast cancer. Deaths from unrelated causes will be censored.
5-Year Distant Recurrence-Free Survival (DRFS) | secondary outcome is calculated from the date of surgery to the time the first event occurs, or if the event is not reported on the last follow-up date.(After 5 years of follow-up observation of subject registration)
  Events for DRFS are defined as the first occurrence of distant recurrence. Local recurrence and contralateral breast cancer will be censored.
5-Year Locoregional Recurrence-Free Survival (LRFS) | secondary outcome is calculated from the date of surgery to the time the first event occurs, or if the event is not reported on the last follow-up date.(After 5 years of follow-up observation of subject registration)
  Events for LRFS include the first occurrence of local or regional recurrence. Distant recurrence and contralateral breast cancer will be censored.
5-Year Nipple Recurrence Rate (NR) | secondary outcome is calculated from the date of surgery to the time the first event occurs, or if the event is not reported on the last follow-up date.(After 5 years of follow-up observation of subject registration)
  NR is defined as the first recurrence of the nipple-areola complex (NAC). Recurrence in the ipsilateral breast or chest muscles, chest wall, regional lymph nodes, contralateral breast, or distant sites will be censored.
Positive Margin Rate (at Surgery) | secondary outcome is calculated from the date of surgery to the time the first event occurs, or if the event is not reported on the last follow-up date.(After 5 years of follow-up observation of subject registration)
  A positive margin is defined as tumor involvement of the NAC, superficial, posterior, or circumferential margins confirmed in the final pathology report. The overall positive margin rate will be analyzed.
Conversion Rate to Open Surgery (RNSM Group Only; at Surgery) | secondary outcome is calculated from the date of surgery to the time the first event occurs, or if the event is not reported on the last follow-up date.(After 5 years of follow-up observation of subject registration)
  In the RNSM group, intraoperative conversion from RNSM to CNSM will be analyzed. Reasons for conversion will be documented.
Operation time | secondary outcome is calculated from the date of surgery to the time the first event occurs, or if the event is not reported on the last follow-up date.(After 5 years of follow-up observation of subject registration)
  Total operative time includes both mastectomy and reconstruction. Each component will be measured separately and analyzed.
30-Day Postoperative Complication Rate | secondary outcome is calculated from the date of surgery to the time the first event occurs, or if the event is not reported on the last follow-up date.(After 5 years of follow-up observation of subject registration)
  The complication rate within 30 days post-surgery will be calculated as the total number of complications per patient in each group. Both the total number of complications per patient and the number of Clavien-Dindo grade III or higher complications per patient will be analyzed. NAC necrosis rate will also be evaluated.
Clavien-Dindo Classification of Postoperative Complications (within 180 days) | secondary outcome is calculated from the date of surgery to the time the first event occurs, or if the event is not reported on the last follow-up date.(After 5 years of follow-up observation of subject registration)
  Postoperative complications will be assessed using the Clavien-Dindo classification. Grade III or higher complications, including flap or implant loss, will be analyzed.
Flap or Implant Loss Rate (within 1 year postoperatively) | Flap or implant loss within 1 year of surgery will be recorded and analyzed.
Patient-Reported Outcomes (between 3 and 12 months postoperatively) | secondary outcome is calculated from the date of surgery to the time the first event occurs, or if the event is not reported on the last follow-up date.(After 5 years of follow-up observation of subject registration)
  Breast satisfaction will be evaluated using the BREAST-Q version 2.0 scale administered before and after mastectomy. Higher scores indicate better outcomes.
Surgeon Satisfaction (between 3 and 12 months postoperatively) | secondary outcome is calculated from the date of surgery to the time the first event occurs, or if the event is not reported on the last follow-up date.(After 5 years of follow-up observation of subject registration)
  Surgical satisfaction will be evaluated by the operating surgeon. Overall symmetry, postoperative scarring, and NAC symmetry will be scored using a 0-10 scale, with higher scores indicating better outcomes.
  Overall symmetry, postoperative scar, and NAC symmetry are measured using scoring system 0-10. The higher scores are, the better an outcome is.
Cost-Effectiveness (between 3 and 12 months postoperatively; optional) | secondary outcome is calculated from the date of surgery to the time the first event occurs, or if the event is not reported on the last follow-up date.(After 5 years of follow-up observation of subject registration)
  Cost-effectiveness will be assessed between 3 and 12 months after the final surgery using the Korean version of the EuroQol 5-Dimension (EQ-5D) questionnaire. Higher scores indicate better outcomes across all dimensions.
30-Day Estimated Postoperative Complication Rate | secondary outcome is calculated from the date of surgery to the time the first event occurs, or if the event is not reported on the last follow-up date.(After 5 years of follow-up observation of subject registration)
  Based on a sample size of 790 (632 after accounting for 20% dropout), the study has at least 80% power to detect various assumed complication rates between the conventional and robotic groups, with a non-inferiority margin of 7.5%. The assumed 30-day complication rate for the conventional group is 25-50%. The maximum 30-day complication rate for the robotic group to be considered non-inferior is presented in Table 2. These will be analyzed as secondary endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Seok Park, MD, PhD, Principal Investigator — Yonsei University
Locations (17):
- South Korea (17):
  - Samsung Changwon Medical Center, Changwon
  - Keimyung University Dongsan Hospital, Daegu
  - Kyungpook National University Chilgok Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Myongji Hospital, Goyang-si
  - The Catholic University of Korea, Incheon ST. Mary's Hospital, Incheon
  - Kosin University Gospel Hospital, Pusan
  - Chungnam National University Sejong Hospital, Sejong
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Ansan Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Soonchunhyang University Hospital Seoul, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul
  - Yongin Severance Hospital, Yongin-si

IPD SHARING:
Plan to Share IPD: No